CLINICAL TRIAL: NCT00688909
Title: Open-label, Single-arm, Multicenter Study to Evaluate the Rheumatological Tolerability of Letrozole as an Adjuvant Breast Cancer Treatment in Postmenopausal Women Who Are Intolerant and Discontinue Anastrozole Due to Grade 2-3 Arthralgia-myalgia
Brief Title: Rheumatological Evaluation of Anastrozole and Letrozole as Adjuvant Treatment in Post-menopausal Women With Breast Cancer
Acronym: REAL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CFEM345DUS59
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2021-05-24 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
Keywords: breast cancer; adjuvant treatment in post menopausal women; letrozole; arthralgia-myalgia
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Letrozole (Experimental): Participants received 2.5 milligram (mg) of Letrozole tablets orally once daily (QD) for a period of 24 weeks.
  Interventions: Drug: letrozole

INTERVENTIONS:
Drug: letrozole — 2.5 mg daily by mouth for 6 months
  Other Names: Femara

SUMMARY:
This study will evaluate whether patients who are intolerant and discontinue anastrozole due to grade 2-3 arthralgia-myalgia have a decrease in rheumatological symptoms while taking letrozole

DETAILED DESCRIPTION:
This is a multi-center prospective non-randomized single arm, open label trial in postmenopausal HR positive early breast cancer patients who experience grade 2-3 arthralgia-myalgia while on anastrozole, resulting in the discontinuation of anastrozole. After a 2-3 week period without any aromatase inhibitor treatment, eligible patients will initiate letrozole treatment at a dose of 2.5mg per day for a duration of 24 weeks. If a patient has breast cancer recurrence or is intolerant to letrozole during the 24 week period, the drug will be discontinued.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women with HR+ early stage breast cancer at the time of initial diagnosis. For study purposes, postmenopausal is defined as:

   * Age ≥ 50 y and amenorrheic for 12 or more months.
   * Age ≥ 50 y and amenorrheic for 3 or more months after receiving adjuvant chemotherapy.
   * Age < 50 y and amenorrheic for 12 or more months.
   * Prior bilateral oophorectomy.
   * Prior hysterectomy and has postmenopausal levels of FSH, LH, and estradiol as per local institutional standards.
   * Age > 55 y and prior hysterectomy.
2. Patients who are intolerant and discontinue anastrozole 2-3 weeks prior to study entry when given as adjuvant treatment for HR+ early stage breast cancer due to grade 2-3 (NCI-CTCAE V3) arthralgia-myalgia.
3. Hormone receptor-positive tumors as defined by institutional standards.
4. ECOG performance status of 0, 1, or 2
5. Consent to participate in the trial. -

Exclusion Criteria:

1. Postmenopausal women with HR+ metastatic or locally relapsed breast cancer excluding chest wall recurrence with no evidence of systemic disease.
2. Recent history of pain associated with non-traumatic bone fracture.
3. Pain requiring chronic use of analgesics (due to any reason).
4. History of rheumatological disease except osteoarthritis.
5. Prior hormonal therapy with AIs other than anastrozole.
6. Systemic hormone replacement therapy (HRT) less than 4 weeks before study entry other than Estring®, Vagifem® or low dose estrogen vaginal cream.
7. Concomitant disease which significantly affects quality of life.
8. Patient unable to complete self administered questionnaire.
9. Patients unable to sign consent form.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2008-03; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (48):
- United States (48):
  - Clearview Cancer Center, Huntsville, Alabama
  - Hematology Oncology Services of Arkansas, Little Rock, Arkansas
  - Grass Valley Hematology Oncology, Grass Valley, California
  - Aptium Oncology - Comprehensive Cancer Care of the Desert, Palm Springs, California
  - Bay Area Cancer Research Group, Pleasant Hill, California
  - Front Range Specialist, Fort Collins, Colorado
  - Lynn Cancer Center, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Memorial Cancer Center, Hollywood, Florida
  - Palm Beach Cancer Specialists, West Palm Beach, Florida
  - Northeast Georgia Cancer Care, LLC, Athens, Georgia
  - Augusta Oncology, Augusta, Georgia
  - Oncology Specialist of North Georgia, Gainesville, Georgia
  - The Cancer Instiute at Alexian Brothers, Elk Grove Village, Illinois
  - Evanston Northwestern Hospital, Evanston, Illinois
  - Edward H. Kaplan MD & Associates - North Shore Cancer Research Associates, Skokie, Illinois
  - Cancer Care of Kansas, Wichita, Kansas
  - Kentuckiana Cancer Institute, Louisville, Kentucky
  - Mercy Hospital, Portland, Maine
  - Mercey Hospital, Baltimore, Maryland
  - Maryland Hematology Oncology Associates, PA, Baltimore, Maryland
  - Suburban Hospital Cancer Program, Bethesda, Maryland
  - Hematology Oncology Asssociates of Ohio & Michigan, Lambertville, Michigan
  - Center for Cancer Care and Research, St Louis, Missouri
  - Ballas Cancer Center, LLC DBA - St Louis, St Louis, Missouri
  - Southeast Nebraska Hematology & Oncology Consultants, Lincoln, Nebraska
  - Trinitas Comprehensive Cancer Center, Elizabeth, New Jersey
  - Hematology-Oncology Assoc of Northern New Jersey, Morristown, New Jersey
  - Somerset Hematology & Oncology, Somerville, New Jersey
  - Cooper University Hospital, Voorhees Township, New Jersey
  - Broom Oncology, Binghamton, New York
  - Cancer Care of W. NC, Asheville, North Carolina
  - Marion L. Shepard Cancer Center, Washington, North Carolina
  - Summa Health System, Akron, Ohio
  - Mukesh Bhatt, MD, INC., Medina, Ohio
  - Berks Hematology Oncology, West Reading, Pennsylvania
  - South Carolina Oncology Associates, Columbia, South Carolina
  - The West Clinic, Memphis, Tennessee
  - Tenessee Oncology, Nashville, Tennessee
  - Coastal Bend Cancer Center, Corpus Christi, Texas
  - Center for Oncology Research and Treatment, Dallas, Texas
  - Central Utah Clinic, American Fork, Utah
  - Northern Utah Associates, Ogden, Utah
  - Medical Oncology & Hematology Associates of Northern Virginia, Fairfax, Virginia
  - Rockingham Memorial Hospital Regional Cancer Center, Harrisonburg, Virginia
  - Peninsula Cancer Center, Newport News, Virginia
  - Green Bay Oncologist, St Vincent Hospital, Green Bay, Wisconsin
  - Oncology Alliance, Wauwatosa, Wisconsin

REFERENCES:
- See also: Results for CFEM345DUS59 from the Novartis Clinical Trials Results Database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=3500

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled 261 participants at 45 centers in United States.
Pre-assignment Details: It was estimated it would be necessary to enroll 228 patients so that the percentage of patients discontinuing due to arthralgia-myalgias would be 50%, within 6.5% of the true percentage with 95% confidence.
Period: Overall Study
Arm/Group | Letrozole
Started | 261
Completed | 228
Not Completed | 33
Not completed — Adverse Event | 28
Not completed — Patient withdrew consent | 2
Not completed — Administrative problems | 1
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Letrozole
Number analyzed (Participants) | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (10.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 261
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 235
  Black | 14
  Asian | 3
  Other | 9
Relevant Medical and Surgical History [Count of Participants; unit: Participants]
  Yes | 261
  No | 0
Rheumatology History [Count of Participants; unit: Participants]
  Yes | 261
  No | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Discontinuing Due to Grade 2 or Higher Arthralgia-myalgia.
Description: The arthralgia status and the myalgia status were separately graded at Baseline (V1), Week 12 (V3) , and Week 24/EOS (V4). The grades of 0 for no pain, 1 for mild pain, 2 for moderate pain, 3 for severe pain, and 4 for disabling pain were used.
Time Frame: End of Study (24 weeks)
Population: Safety set: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole
Number analyzed (Participants) | 261
Participants | 25

2. Secondary Outcome: Time to Discontinuation Due to Grade 2 or Higher Arthralgia- Myalgia.
Description: For patients who discontinued from the study due to either grade 2 or higher arthralgia-myalgia, the time to discontinuation was calculated as the duration between the Visit 1 date and the last dose date. If the last dose date was missing, the EOS date was used.
Time Frame: End of Study (24 weeks)
Population: Safety set: All participants who received at least one dose of study drug.
Measure: Mean (Standard Error); unit: days
Arm/Group | Letrozole
Number analyzed (Participants) | 261
days | 156.98 (1.94)

3. Secondary Outcome: Percentage of Participants Discontinuing, Irrespective of Cause
Description: The percentage of patients who discontinued from the study irrespective of the reasons.
Time Frame: End of Study (24 weeks)
Population: Safety set: All participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Letrozole
Number analyzed (Participants) | 261
Participants | 33

4. Secondary Outcome: Change in Brief Pain Inventory (BPI) Composite Score
Description: The BPI is a pain assessment tool for use with cancer patients. The BPI measures both the intensity of pain (sensory dimension) and interference of pain in the patient's life (reactive dimension). It also queries the patient about pain relief, pain quality, and patient perception of the cause of pain. The BPI composite score was calculated based on questions 3 to 6 of the BPI Questionnaire (short form). First each question was scored from 0 (no pain) to 10 (pain as bad as you can imagine) and circled on the CRF. Then a composite score was calculated as the mean of the scores. If any answer was missing, the composite score was set to missing. Change in BPI composite score indicates the change from baseline at week 24.
Time Frame: Baseline, 24 weeks (End of Study)
Population: Safety set: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Letrozole
Number analyzed (Participants) | 261
score on a scale
  Baseline visit: number analyzed (Participants) | 257
  Baseline visit | 2.78 (2.00)
  Week 24: number analyzed (Participants) | 243
  Week 24 | -0.46 (2.09)

5. Secondary Outcome: Change in Disability Index as Assessed by Health Assessment Questionnaire (HAQ)
Description: The HAQ is a validated, patient-oriented outcome assessment instrument. The short version '2 page HAQ' was used. It contains the HAQ Disability Index (HAQ-DI), the HAQ visual analog scale (VAS) for pain and the VAS patient global health scale. The Stanford HAQ 20-item disability scale was utilized for scoring of the Disability Index. The items were first scored within each category with values 0 to 3 (0 = Without any difficulty, 1 = With some difficulty, 2 = With much difficulty, 3 = Unable to do). The score for the disability index was the mean of the eight category scores. If more than 2 of the 8 categories, or >25%, were missing, the scale was not scored. If ≤2 of the categories were missing, the sum of the categories was divided by the number of answered categories. Change in Disability Index indicates the change from baseline at week 24.
Time Frame: Baseline, Visit 1(24 weeks = End of Study)
Population: Safety set: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Letrozole
Number analyzed (Participants) | 261
score on a scale
  Visit 1 (Baseline visit): number analyzed (Participants) | 260
  Visit 1 (Baseline visit) | 0.54 (0.55)
  Visit 4 (Week 24): number analyzed (Participants) | 252
  Visit 4 (Week 24) | -0.07 (0.47)

6. Secondary Outcome: Change in Pain as Assessed by Visual Analog Scale (VAS) Scale of the Health Assessment Questionnaire (HAQ)
Description: The HAQ is a validated, patient-oriented outcome assessment instrument. The short version '2 page HAQ' was used. It contains the HAQ Disability Index (HAQ-DI), the HAQ visual analog scale (VAS) for pain and the VAS patient global health scale. The VAS is a tool used to help a person rate the intensity of certain sensations and feelings, such as pain. The visual analog scale for pain is a straight line with one end meaning no pain and the other end meaning the worst pain imaginable. For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [100-mm scale]). A higher score indicates greater pain intensity. Change in pain as assessed by VAS indicates the change from baseline at week 24.
Time Frame: Baseline, Visit 1 (24 weeks = End of Study)
Population: Safety set: All participants who received at least one dose of study drug.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Letrozole
Number analyzed (Participants) | 261
score on a scale
  Visit 1 (Baseline visit): number analyzed (Participants) | 255
  Visit 1 (Baseline visit) | 28.9 (24.22)
  Visit 4 (Week 24): number analyzed (Participants) | 245
  Visit 4 (Week 24) | -6.4 (29.30)

ADVERSE EVENTS:
Time Frame: Adverse events were collected From Start of the Study up to EOS (Week 24)
Description: Safety set: All participants who received at least one dose of study drug.
Groups:
- Letrozole 2.5 mg: Participants received 2.5 milligram (mg) of Letrozole tablets orally once daily (QD) for a period of 24 weeks.
Arm/Group | Letrozole 2.5 mg
All-Cause Mortality (participants affected / at risk) | 0/261
Serious Adverse Events (participants affected / at risk) | 5/261
Other Adverse Events (participants affected / at risk) | 163/261
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole 2.5 mg (N=261)
Cholecystitis chronic (Hepatobiliary disorders) | 1
Post procedural bile leak (Injury, poisoning and procedural complications) | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Mania (Psychiatric disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Letrozole 2.5 mg (N=261)
Constipation (Gastrointestinal disorders) | 8
Diarrhoea (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 13
Fatigue (General disorders) | 32
Oedema peripheral (General disorders) | 10
Sinusitis (Infections and infestations) | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 88
Myalgia (Musculoskeletal and connective tissue disorders) | 78
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 8
Depression (Psychiatric disorders) | 13
Insomnia (Psychiatric disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 6
Hot flush (Vascular disorders) | 37
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No